CLINICAL TRIAL: NCT07398495
Title: Effects of Multimodal Training on Muscle Function and Glucose Metabolism in Middle-Aged and Older Adults With Type 2 Diabetes Mellitus and Sarcopenia
Brief Title: Multimodal Training Effects in Middle-Aged and Older Adults With Diabetic Sarcopenia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Principal Investigator, yueh chu wu, Diabetes Educator, Chung Shan Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CSH-2026-A-036
Record Dates: First submitted 2026-02-04; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Type 2 Diabetes Mellitus (T2DM); Sarcopenia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Sarcopenia | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Multimodal Exercise) (Experimental): • Arm Description: Participants in this group will engage in a 12-week multimodal exercise program. The program includes supervised training sessions, home-based exercises, and digital support. They will also receive a "Diabetes and Muscle Health Handbook" to guide their training.
  Interventions: Behavioral: Multimodal Exercise Program
- Control Group (Standard Care) (No Intervention): Participants in this group will serve as the control. They will receive a "Nutrition and Muscle Health Education Sheet" at the beginning of the study. They will not participate in the multimodal exercise program and will continue with their routine health management based on existing medical advice.

INTERVENTIONS:
Behavioral: Multimodal Exercise Program — Participants will engage in a 12-week multimodal exercise program comprising supervised training sessions, home-based exercises, and digital support. To facilitate adherence and proper technique, participants will also receive a "Diabetes and Muscle Health Handbook" as a training guide.
  Other Names: Control Group
  Arms: Intervention Group (Multimodal Exercise)

SUMMARY:
This study aims to investigate the effects of a 12-week multimodal exercise intervention on middle-aged and older adults (aged 45~85 years) with Type 2 Diabetes Mellitus (T2DM). The program combines supervised training, home-based sessions, and digital support to improve muscle function, physical performance, metabolic control, and quality of life.

DETAILED DESCRIPTION:
Middle-aged and older adults with T2DM, particularly in Asian populations, face a heightened risk of sarcopenia. This condition leads to a decline in muscle mass and function, negatively impacting quality of life. Effective interventions are urgently needed to slow disease progression. This randomized controlled trial will recruit 58 adults. Participants will be randomly assigned to either a control group or an intervention group. The intervention involves a multimodal exercise program and educational materials, while the control group receives standard health education. Assessments will be conducted at baseline, week 12, and week 24 to evaluate physical function, sarcopenia risk, metabolic control, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with both Type 2 Diabetes Mellitus (T2DM) and sarcopenia.
* Maintained on a stable regimen of oral hypoglycemic agents.
* Aged 45 years or older.
* Capable of communicating effectively in Mandarin or Taiwanese.
* Willing to provide informed consent or have it obtained from a legally authorized representative.

Exclusion Criteria:

* • Limited limb or joint function that prevents exercise (e.g., recent fractures or dislocations).

  * Communication barriers or severe emotional/psychological issues (e.g., uncontrolled depression or severe mental illness).
  * Severe cognitive impairment (e.g., dementia).
  * End-stage renal disease (ESRD).
  * Major comorbidities or complications, including active diabetic foot ulcers, amputation, recent myocardial infarction, severe autonomic neuropathy, or a history of stroke within the last 3 years.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2026-03-02 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Physical Function (5TSTS) | Change from Baseline at Week 12 and Week 24
  The Five-Times Sit-to-Stand Test (5TSTS) assesses lower limb muscle power. Participants are asked to stand up and sit down five times as quickly as possible with arms folded. The time to completion is recorded in seconds and analyzed as a continuous variable. Longer completion times indicate poorer physical performance
Handgrip Strength (HGS) | Change from Baseline at Week 12 and Week 24
  Measured using a digital dynamometer (e.g., Jamar or equivalent). Participants perform the test in a standing position with the arm fully extended. Two trials are performed for each hand, and the highest value (kg) is used for analysis. Low muscle strength is defined according to AWGS 2019 criteria (<28 kg for men and <18 kg for women).
Skeletal Muscle Mass Index (SMI) | Change from Baseline at Week 12 and Week 24
  Determined by bioelectrical impedance analysis (BIA). Appendicular skeletal muscle mass (ASM, kg) is calculated as the sum of lean mass from both arms and legs. SMI is expressed as ASM divided by height squared (kg/m²). Low muscle mass is defined according to AWGS 2019 cut-off values (<7.0 kg/m² for men and <5.7 kg/m² for women).
Sarcopenia Risk (SARC-CalF) | Change from Baseline at Week 12 and Week 24
  Assessed using the SARC-CalF questionnaire, combining the SARC-F (5 items: strength, walking, rising, climbing stairs, falls; scored 0-10) with calf circumference measurement. Calf circumference ≤34 cm (men) or ≤33 cm (women) adds 10 points to the score. A total SARC-CalF score ≥11 indicates a high risk of sarcopenia.

SECONDARY OUTCOMES:
Glycated Hemoglobin (HbA1c) | Change from Baseline at Week 12 and Week 24
  Metabolic control evaluated by HbA1c levels. Venous blood samples are collected after an overnight fast and analyzed using standardized high-performance liquid chromatography (HPLC). Values are reported as percentages.
Quality of Life (SF-12) | Change from Baseline at Week 12 and Week 24
  Assessed using the 12-Item Short Form Health Survey (SF-12). The survey covers eight domains summarized into two composite scores: the Physical Component Summary (PCS) and the Mental Component Summary (MCS). Scores range from 0 to 100, with higher scores indicating better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Chung Shan Medical University Hospital, Taichung, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No